CLINICAL TRIAL: NCT05313360
Title: The Association Between Sarcopenia and Urinary Incontinence and the Effect of Physical Activity Among Over 50 Years Old Adults in South-Danubia
Brief Title: Association Between Sarcopenia and Urinary Incontinence And Effect Of Physical Activity Among Over 50 Years Old Adults
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 9080 - PTE 2021
Record Dates: First submitted 2022-01-06; First posted 2022-04-06 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Urinary Incontinence; Sarcopenia
Keywords: Urinary Incontinence; Sarcopenia
MeSH Terms: conditions — Urinary Incontinence; Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As far as the investigators know, until this moment no research has investigated the prevalence of Sarcopenia in both sexes in Hungary. Additionally, no research discovered the association between sarcopenia and UI and the effect of physical activity level on these geriatric conditions in Hungary.

Furthermore, it is known that Sarcopenia and UI are causing negative psychological, physical, and social effects on the geriatrics who are suffering from these conditions, not to mention the increase in health care costs. In an attempt to decrease these negative effects, there is a need for a deeper understanding of these conditions by identifying the relationship between them and understanding the risk factors that might cause them. The finding of this study would help with determining those risk factors that are causing these geriatric conditions (Sarcopenia and UI).

Last, this study will provide accurate numbers and statistics to the Hungarian health organizations and educational institutions about the prevalence of sarcopenia and UI which will help shed the light on the importance of these problems among older adults in Hungary.

This Cross-sectional study aim to:

1. Explore and study physical activity levels among aging adults of both sexes in Hungary.
2. To determine the prevalence of sarcopenia and UI among elderly individuals in Hungary.
3. Investigate the associations between sarcopenia and urinary incontinence among older adults (≥ 50 years).
4. Identify the effect of physical activity level on the occurrence of Sarcopenia and Urinary incontinence

Hypothesis:

1. The investigators hypothesize that sarcopenia is a risk factor to have UI.
2. The investigators hypothesize that reduced physical activity level is also associated with sarcopenia and/or UI.

ELIGIBILITY:
Inclusion Criteria:

• Any person who is 50 years old or older

Exclusion Criteria:

• Individuals who cannot provide reliable clinical information due to cognitive disorders.

Individuals who are having any neurodegenerative disorders (E.g; Parkinson).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is any participant who is 50 years or older, and living in the South Danubia region, in Hungary.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Sarcopenia and urinary incontinence | Day 1
  Investigate the associations between sarcopenia and urinary incontinence among older adults (≥ 50 years).
Physical activity level effect | Day 1
  Identify the effect of Physical activity level on the occurrence of Sarcopenia and Urinary incontinence.

SECONDARY OUTCOMES:
Prevalence of Sarcopenia and Urinary incontinence | Day 1
  To determine the prevalence of sarcopenia and UI among elderly individuals in Hungary
insights into physical activity levels | Day 1
  Explore and study physical activity levels among aging adults of both sexes in Hungary

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Debes WA, Sadaqa M, Acs P, Kovacs K, Premusz V, Hock M. Sarcopenia risk as a predictor of urinary incontinence in women aged 50 and older: a cross-sectional analysis. Sci Rep. 2025 Jul 26;15(1):27288. doi: 10.1038/s41598-025-11963-2. PMID 40715321